CLINICAL TRIAL: NCT02939040
Title: A Pilot Study of a Brief Pre-Operative Intervention for Patients Undergoing Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Afton Hassett, Psy.D., Associate Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00114087; UMCC 2016.036 (Other: University of Michigan Cancer Center)
Record Dates: First submitted 2016-08-01; First posted 2016-10-19 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: positive activities intervention; peri-operative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Activities Intervention (Experimental): Patients will note at least one positive event each day, write it down on a slip of paper and then deposit this piece of paper in a piggy bank. After approximately 21 days, the participant reads each one the night before surgery.
  Interventions: Behavioral: Positive Activities
- Usual Care Group (No Intervention): The control group will serve to show the relative benefits of the Positive Piggy Bank intervention. These participants will follow the same questionnaire completion procedures.

INTERVENTIONS:
Behavioral: Positive Activities — The PPB intervention involves noting at least one positive event each day, writing it down on a slip of paper and then depositing this piece of paper in a piggy bank. This practice is to take place at the end of the day, every day over a circumscribed period of time. At the end of the "deposit period" the participant "closes the account" and makes a full withdrawal by taking all of the slips out of the piggy bank and reading each one the night before surgery.
  Arms: Positive Activities Intervention

SUMMARY:
This study is to assess the feasibility of using a positive activities intervention, Positive Piggy Bank, in newly diagnosed women with breast cancer who will soon undergo surgery. A randomized controlled pilot trial of a brief self-guided positive activities intervention, The Positive Piggy Bank (PPB), compared to Treatment as Usual. The PPB intervention involves noting at least one positive event each day, writing it down on a slip of paper and then depositing this piece of paper in a piggy bank. This practice is to take place at the end of the day, every day over a circumscribed period of time. At the end of the "deposit period," in the case of this study after approximately 21 days, the participant "closes the account" and makes a full withdrawal by taking all of the slips out of the piggy bank and reading each one on the night before surgery.

DETAILED DESCRIPTION:
Fifty participants will complete questionnaires at baseline (Day 1), then they will be randomized 1:1 to the Positive Piggy Bank condition (n=25) or Treatment as Usual (n = 25) approximately 3 weeks before surgery. Post-intervention (Day of Surgery) and 14 days post-surgery, participants will complete the same questionnaires. The 14 day post surgery questionnaires will be administered by phone.

Intervention Procedures - The Positive Piggy Bank. Participants randomized to this group will first get an overview of the intervention, learn about the rationale for this treatment, and receive supplies including the instructions on a decorative card, a piggy bank, and paper currency slips (pieces of lined paper with a place for the date). Participants in this group will be instructed to do the activities as detailed above in the Positive Piggy Bank instructions daily until the evening before surgery (approximately 21 days). On the evening before surgery, they are to "close their account" by opening the piggy bank and reviewing all of the slips of paper.

Study personnel will contact patients within 72 hours of beginning the study to answer questions and/or provide encouragement. Participants will also be contacted on the day before surgery to let them know that they should read all of their currency slips and reminded to bring their currency slips with them to the hospital on the day of surgery.

On the day of surgery, prior to surgery they will complete the first set of follow-up questionnaires. They will also be reminded that these same follow-up questionnaires will be administered by phone 14 days after surgery.

The control group will serve to show the relative benefits of the Positive Piggy Bank intervention. These participants will follow the same questionnaire completion procedures as listed above including phone calls. The phone call at 72 hours will be to simply thank them for their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Recent diagnosis of breast cancer with pending surgery as primary treatment for breast cancer.
2. Ages 18 and above.
3. Able to read/understand English and give consent.
4. Willing and able to comply with all aspects of study procedures.
5. No plan to initiate a new program that could affect well-being during the study period (e.g., psychotherapy, new exercise regimen, meditation classes).

Exclusion Criteria:

1. Planned neoadjuvant systemic therapy.
2. Having a psychotic disorder or the presence of another psychiatric condition (e.g., severe depression [i.e., score on the PHQ-9], suicidal ideation) or cognitive impairment (e.g., severe dyslexia, traumatic brain injury) limiting ability to give consent and/or participate fully in the study.
3. Other factors that at the discretion of the investigators would adversely affect study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a Positive Activities Intervention | Day 1 (baseline), Day of Surgery and 14 Days Post Surgery
  The primary objective of this study is to assess the feasibility of using a positive activities intervention, Positive Piggy Bank, in newly diagnosed women with breast cancer who will soon undergo surgery. We will also explore changes in subjective well-being and post-surgical symptoms in response to the intervention in order to power a larger trial.

SECONDARY OUTCOMES:
Symptom Burden | Day 1 (baseline), Day of Surgery and 14 Days Post Surgery
  Measured by the MSAS
Fatigue | Day 1 (baseline), Day of Surgery and 14 Days Post Surgery
  Measured by the PROMIS Profile 29
Sleep | Day 1 (baseline), Day of Surgery and 14 Days Post Surgery
  Measured by the PROMIS Profile 29
Depressive Symptoms | Day 1 (baseline) to 14 Days Post Surgery
  Measured by the PROMIS Profile 29
Social Roles | Day 1 (baseline), Day of Surgery and 14 Days Post Surgery
  Measured by the PROMIS Profile 29

CONTACTS AND LOCATIONS:
Overall Officials: Afton Hassett, Psy.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Chronic Pain and Fatigue Research Center, Ann Arbor, Michigan, United States